CLINICAL TRIAL: NCT00362271
Title: Effects of Aripiprazole on the Steady-State Pharmacokinetics of Venlafaxine in Healthy Subjects
Brief Title: Aripiprazole and Effexor XR Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CN138-462 ST
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — Aripiprazole

ARMS (1):
- 1 (Other)
  Interventions: Drug: Venlafaxine on Day -4 to day 14, Aripiprazole dosed starting on Day 1: 3 days at 10 mg, 4 days at 1 mg and 7 days at 20 mg.

INTERVENTIONS:
Drug: Venlafaxine on Day -4 to day 14, Aripiprazole dosed starting on Day 1: 3 days at 10 mg, 4 days at 1 mg and 7 days at 20 mg. — Tablets, Oral, Venlafaxine: 75 mg; Aripiprazole: 10, 15, 20 mg once daily, 14 days.
  Other Names: Abilify

SUMMARY:
The purpose of this clinical research study is to learn whether aripiprazole has effect on the steady-state pharmacokinetics of venlafaxine in healthy subjects. The safety and tolerability of aripiprazole and venlafaxine co-administration will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, ages 18 to 45 (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized.
* Body Mass Index (BMI) of 18 to 33 kg/m2, inclusive.

Exclusion Criteria:

* Subjects with a decrease in SBP of >=20 mm Hg and increase in HR of >=20 bpm after 2 minutes standing vs. 2 minutes supine at screening or with frank orthostatic hypotension at screening.
* Supine BP of 90/50 mm Hg or lower at screening
* SBP >=140 mm Hg or DBP >=90 mm Hg at screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Multiple dose PK parameters for venlafaxine+metabolite when administered alone and with aripiprazole will be derived. Cmin for aripiprazole,dehydro-aripiprazole will be measured

SECONDARY OUTCOMES:
Safety will be based on review of AEs, VS, ECGs, physical exam, clinical labs

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Miami, Florida, United States

REFERENCES:
- [Derived] Boulton DW, Balch AH, Royzman K, Patel CG, Berman RM, Mallikaarjun S, Reeves RA. The pharmacokinetics of standard antidepressants with aripiprazole as adjunctive therapy: studies in healthy subjects and in patients with major depressive disorder. J Psychopharmacol. 2010 Apr;24(4):537-46. doi: 10.1177/0269881108096522. Epub 2008 Oct 2. PMID 18832427